CLINICAL TRIAL: NCT03160209
Title: LCCC 1608 - HIV and Other Risk Factors for Esophageal Squamous Cell Carcinoma in Malawi
Brief Title: HIV and Other Risk Factors for Esophageal Squamous Cell Carcinoma in Malawi
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 1608
Record Dates: First submitted 2017-05-04; First posted 2017-05-19 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: risk factors; case-control study
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 300 esophageal cases: diagnosed with histologically confirmed ESCC
- 300 patient controls: without a history of esophageal cancer or esophageal squamous dysplasia, a history of other cancer, or upper gastrointestinal diseases

SUMMARY:
The primary purpose of this single-center, case-control, non-interventional study is to determine risk factors which contribute to the development of esophageal squamous cell carcinoma (ESCC) at Kamuzu Central Hospital (KCH) and St. Gabriel Hospital (SGH) in Malawi.

DETAILED DESCRIPTION:
RATIONALE FOR RESEARCH

The Rift Valley of Africa is a 'hot spot' for ESCC, yet little is known about the etiology of this disease in Sub-Saharan Africa. In Malawi, ESCC is the third commonest cancer nationwide behind Kaposi sarcoma and cervical carcinoma. Among cancers that are not classically HIV-related, ESCC has the highest incidence in Malawi. The ESCC burden recorded in the national cancer registry is also likely an underestimate, as many cases may go undiagnosed and unregistered. Additionally, few data are available on the epidemiology of ESCC in Malawi, and underlying reasons for high frequency of the disease are largely unknown. This knowledge gap is a major barrier to public health prevention efforts. Given that survival after ESCC diagnosis is dismal in Malawi (12% at 1 year), developing evidence-based prevention efforts is paramount.

The proposed study will make a significant contribution to existing literature from Malawi and Sub-Saharan Africa in several important respects. First, previous epidemiologic studies of ESCC in Malawi have been limited by challenges with appropriate control selection, which may have limited the validity of their findings. Secondly, our study will include prospective clinical follow-up of confirmed ESCC cases as they receive treatment under local conditions to provide accurate survival estimates. Thirdly, biospecimens from consenting patients will permit etiology and pathogenesis studies to understand mechanisms of ESCC development, which can be correlated with high-quality clinical and epidemiologic data. Finally, we plan to coordinate with other ESCC researchers in eastern and southern Africa to harmonize data collection, and help create a regional consortium in which Malawi can be a founding member and active participant.

Primary Objective: Identify demographic and environmental risk factors for ESCC through a case-control study implemented at KCH and SGH. Hypothesis: Modifiable risk factors contribute significantly to ESCC. These include polycyclic aromatic hydrocarbon (PAH) exposure from various sources, excessively hot beverages, dietary factors such as maize fumonisin and low selenium, and HIV infection.

Secondary Objective: Identify common genetic and epigenetic alterations in germline and somatic DNA associated with ESCC development. Hypothesis: Recurring genetic and epigenetic alterations can facilitate risk stratification, development of early detection biomarkers, and identification of novel treatment strategies.

Procedures

After informed consent and study enrollment, subjects will be interviewed using a structured questionnaire and provide biological samples including saliva, blood, urine, and toenail clippings. Esophageal biopsies will be taken for diagnostic confirmation and to support molecular studies. If patients suspected to have ESCC are enrolled but then pathologically confirmed to have an alternate diagnosis, they will be withdrawn. HIV testing will be offered to all participants, and CD4, HIV RNA, and ART status documented for HIV-infected participants. Exposures will be measured using the questionnaire and laboratory analyses of saliva, blood, urine, and toenail samples. We will collect information on: demographic characteristics; HIV status; tobacco and drug use; alcohol consumption; medical history; family history of cancer; indoor air pollution; occupational history; diet, cooking, and food preservation; beverage history including temperature; farming; signs and symptoms of upper gastrointestinal disease; oral health; anthropometric indices; and reproductive history. To examine correlates with patient outcomes, telephone follow-up to assess vital status will be done every 3 months until 2 years from enrollment. Biological samples will be stored in freezers and transferred to the US only for assays that are currently unavailable in Malawi. Laboratory testing will include serum selenium level, blood and urine testing for PAH exposure, tumor immunohistochemistry assays, salivary DNA isolation for genetic studies, and molecular profiling of ESCC tumors.

Analysis

Sample size will include 300 ESCC cases and 300 controls; 66-68 case control pairs will be enrolled per year, over 3 years, assuming a response rate of 75% in the endoscopy clinic. With 300 case-control pairs, estimated statistical power for an exposure with control population prevalence of 10% and OR 2.0 is 81%, using alpha level 0.05, with higher power for higher control exposure rates and odds ratios. Expected prevalence for key exposures (tobacco and alcohol, hot tea, PAH exposure, selenium deficiency, HIV) is 10-50% in the control population. To assess epidemiologic risk factors for ESCC, we will use logistic regression to estimate odds ratios and 95% confidence intervals for each exposure, while controlling for possible confounders. Survival estimates will be generated using Kaplan-Meyer curves to estimate overall survival at 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Cases Inclusion Criteria

  * All patients > 18 years of age diagnosed with histologically confirmed ESCC are eligible to be a case regardless of sex or place of residence.
  * Diagnosis of ESCC (histologically confirmed)
  * Subject able to understand and provide written consent in English or Chichewa
  * Able to understand and comply with study procedures for the entire length of the study

Controls Inclusion Criteria

* All patients > 18 years of age without a history of esophageal cancer or esophageal squamous dysplasia, a history of other cancer, or upper gastrointestinal diseases are eligible to be controls, regardless of age, sex, or place of residence
* Subject able to understand and provide written consent in English or Chichewa
* Able to understand and comply with study procedures for the entire length of the study

Exclusion Criteria:

* Cases Exclusion Criteria

  * Healthcare provider determines it is unsafe to perform a biopsy
  * Mental impairment which precludes provision of informed consent
  * Patients who are unable to provide their past medical history

Controls Exclusion Criteria

* All patients > 18 years of age with a history of esophageal cancer or esophageal squamous dysplasia, a history of other cancer, or upper gastrointestinal diseases are ineligible to be controls
* Patients with significant difficulty swallowing
* Mental impairment which precludes provision of informed consent
* Patients who are unable to provide their past medical history

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 300 cases diagnosed with histologically confirmed ESCC and 300 patient controls without a history of esophageal cancer or esophageal squamous dysplasia, a history of other cancer, or upper gastrointestinal diseases, 18 years, and older, male/female in Malawi.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Risk factors for ESCC - HIV Infection | 2 years
  To identify risk factors for ESCC through a case-control study implemented at a national teaching hospital, specifically focused on the following exposures: HIV infection, PAH exposure, Dietary factors including fumonisin and selenium, Scalding hot beverages and foods, Tobacco and alcohol consumption
Survival estimates after ESCC diagnosis in Malawi. | 2 years
  To assess survival after ESCC diagnosis in Malawi.
Risk factors for ESCC - HIV Infection | 2 years
  To identify risk factors for ESCC through a case-control study implemented at a national teaching hospital, specifically focused on the following exposures: HIV infection
Risk factors for ESCC - PAH exposure | 2 years
  To identify risk factors for ESCC through a case-control study implemented at a national teaching hospital, specifically focused on the following exposures: PAH exposure
Risk factors for ESCC - Dietary factors including fumonisin and selenium | 2 years
  To identify risk factors for ESCC through a case-control study implemented at a national teaching hospital, specifically focused on the following exposures: Dietary factors including fumonisin and selenium
Risk factors for ESCC - Scalding hot beverages and foods, | 2 years
  To identify risk factors for ESCC through a case-control study implemented at a national teaching hospital, specifically focused on the following exposures: Scalding hot beverages and foods
Risk factors for ESCC - Tobacco and alcohol consumption | 2 years
  To identify risk factors for ESCC through a case-control study implemented at a national teaching hospital, specifically focused on the following exposures: Tobacco and alcohol consumption

SECONDARY OUTCOMES:
The common somatic genetic and epigenetic alterations in ESCC tumors from Malawi. | 2 years
  To identify and characterize common somatic genetic and epigenetic alterations in ESCC tumors from Malawi.
The germline genetic and epigenetic alterations associated with susceptibility to ESCC. | 2 years
  To identify and characterize germline genetic and epigenetic alterations associated with susceptibility to ESCC.

CONTACTS AND LOCATIONS:
Overall Officials: Satish Gopal, MD, MPH, Principal Investigator — UNC-CH
Locations (2):
- Malawi (2):
  - UNC Project, Lighthouse Trust, Lilongwe
  - UNC Project, Lilongwe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu C, Hu Z, He Z, Jia W, Wang F, Zhou Y, Liu Z, Zhan Q, Liu Y, Yu D, Zhai K, Chang J, Qiao Y, Jin G, Liu Z, Shen Y, Guo C, Fu J, Miao X, Tan W, Shen H, Ke Y, Zeng Y, Wu T, Lin D. Genome-wide association study identifies three new susceptibility loci for esophageal squamous-cell carcinoma in Chinese populations. Nat Genet. 2011 Jun 5;43(7):679-84. doi: 10.1038/ng.849. PMID 21642993
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078
- [Background] Metzger R, Schneider PM, Warnecke-Eberz U, Brabender J, Holscher AH. Molecular biology of esophageal cancer. Onkologie. 2004 Apr;27(2):200-6. doi: 10.1159/000076913. PMID 15138356
- [Background] Dlamini Z, Bhoola K. Esophageal cancer in African blacks of Kwazulu Natal, South Africa: an epidemiological brief. Ethn Dis. 2005 Autumn;15(4):786-9. PMID 16259509
- [Background] Mlombe Y, Dzamalala C, Chisi J, Othieno-Abinya N. Oesophageal cancer and Kaposi's sarcoma in Malawi: a comparative analysis. Malawi Med J. 2009 Jun;21(2):66-8. doi: 10.4314/mmj.v21i2.44562. PMID 20345007
- [Background] Msyamboza KP, Dzamalala C, Mdokwe C, Kamiza S, Lemerani M, Dzowela T, Kathyola D. Burden of cancer in Malawi; common types, incidence and trends: national population-based cancer registry. BMC Res Notes. 2012 Mar 16;5:149. doi: 10.1186/1756-0500-5-149. PMID 22424105
- [Background] Munishi MO, Hanisch R, Mapunda O, Ndyetabura T, Ndaro A, Schuz J, Kibiki G, McCormack V. Africa's oesophageal cancer corridor: Do hot beverages contribute? Cancer Causes Control. 2015 Oct;26(10):1477-86. doi: 10.1007/s10552-015-0646-9. Epub 2015 Aug 6. PMID 26245249
- [Background] Kayamba V, Bateman AC, Asombang AW, Shibemba A, Zyambo K, Banda T, Soko R, Kelly P. HIV infection and domestic smoke exposure, but not human papillomavirus, are risk factors for esophageal squamous cell carcinoma in Zambia: a case-control study. Cancer Med. 2015 Apr;4(4):588-95. doi: 10.1002/cam4.434. Epub 2015 Jan 30. PMID 25641622
- [Background] Chen J, Zhang N, Wakai T, Wei L, He Y, Kumagai N, Kitsu K, Wang S, Akazawa K. Effect of the interaction between the amount and duration of alcohol consumption and tobacco smoking on the risk of esophageal cancer: A case-control study. Exp Ther Med. 2010 Nov;1(6):991-997. doi: 10.3892/etm.2010.152. Epub 2010 Sep 29. PMID 22993631
- [Background] Wang JB, Fan JH, Liang H, Li J, Xiao HJ, Wei WQ, Dawsey SM, Qiao YL, Boffetta P. Attributable causes of esophageal cancer incidence and mortality in China. PLoS One. 2012;7(8):e42281. doi: 10.1371/journal.pone.0042281. Epub 2012 Aug 2. PMID 22876312
- [Background] Kumagai N, Wakai T, Akazawa K, Ling Y, Wang S, Shan B, Okuhara Y, Hatakeyama Y, Kataoka H. Heavy alcohol intake is a risk factor for esophageal squamous cell carcinoma among middle-aged men: A case-control and simulation study. Mol Clin Oncol. 2013 Sep;1(5):811-816. doi: 10.3892/mco.2013.142. Epub 2013 Jul 4. PMID 24649251
- [Background] Jessri M, Rashidkhani B, Hajizadeh B, Jessri M, Gotay C. Macronutrients, vitamins and minerals intake and risk of esophageal squamous cell carcinoma: a case-control study in Iran. Nutr J. 2011 Dec 20;10:137. doi: 10.1186/1475-2891-10-137. PMID 22185224
- [Background] Chen Y, Tong Y, Yang C, Gan Y, Sun H, Bi H, Cao S, Yin X, Lu Z. Consumption of hot beverages and foods and the risk of esophageal cancer: a meta-analysis of observational studies. BMC Cancer. 2015 Jun 2;15:449. doi: 10.1186/s12885-015-1185-1. PMID 26031666
- [Background] Sun G, Wang S, Hu X, Su J, Huang T, Yu J, Tang L, Gao W, Wang JS. Fumonisin B1 contamination of home-grown corn in high-risk areas for esophageal and liver cancer in China. Food Addit Contam. 2007 Feb;24(2):181-5. doi: 10.1080/02652030601013471. PMID 17364919